CLINICAL TRIAL: NCT06396130
Title: The Effect of Photobiomodulation Using Low-Level Diode Laser Therapy on Postoperative Pain in Symptomatic Lower Molar Teeth With Irreversible Pulpitis and Apical Periodontitis; a Randomized Controlled Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nour ElGendi, Resident at faculty of dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO 3-3-5 (29/4/24)
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Effect of Photobiomodulation Using Diode Laser

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Photobiomodulation using diode laser (Experimental): Irradiation of periapical tissues with low level diode laser therapy buccally and lingually
  Interventions: Device: Photobiomodulation by low level diode laser
- Placebo/ Mock Laser (Placebo Comparator): Application of laser probe without device activation
  Interventions: Other: Mock Laser Application

INTERVENTIONS:
Device: Photobiomodulation by low level diode laser — Diode laser exposure (Lite Medics 1.00-Watt serial number 148 Ver. SwvM. 150VS108VT.100) will be carried out using a continuous mode with 10 Hz frequency, 980 nm wavelength, and max power 15 WCW. The tip will be applied both at the buccal and the lingual side for 30 s each.
  Arms: Photobiomodulation using diode laser
Other: Mock Laser Application — Placebo for control group
  Arms: Placebo/ Mock Laser

SUMMARY:
this study aims to assess the effect of photobiomodulation using low-level diode laser therapy on postoperative pain after single-visit root canal treatment of mandibular molars with symptomatic irreversible pulpitis and apical periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* . Mature multirooted mandibular molar teeth with: i. Pre-operative sharp pain marked on the VAS scale by reading not less than 6. ii. Clinical diagnosis of symptomatic irreversible pulpitis with periapical periodontitis.

iii. Normal periapical radiographic appearance or slight widening in lamina dura. iv. Positive response and pain provoked by percussion.

- Patients who agree to provide written consent and attend for recall appointments.

Exclusion Criteria:

* Patients who used NSAIDs in the 24 hours before treatment.
* Medically compromised patients having significant systemic disorders. (ASA III or IV).
* Patients with two or more adjacent teeth requiring endodontic treatment.
* Pregnant or nursing females. 5. Teeth that have:

  i. Periodontal affection (with pocket depth greater than 5mm, associated with swelling orfistulous tract, or greater than grade I mobility).

ii. No possible restorability. iii. Signs of pulpal necrosis; associated sinus tract or swelling.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Estimated); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-05-29 (Estimated)

PRIMARY OUTCOMES:
Intensity of postoperative pain | 24, 48 and 72 hours
  Using modified VAS

SECONDARY OUTCOMES:
Total number of analgesic tablets taken in case of intolerable pain | Post instrumentation at 24, 48 and 72 hours
  Counted and recorded by the patient on a special table.